CLINICAL TRIAL: NCT06851260
Title: A Multi-center Prospective Randomized Controlled Study on the Anatomical Relationship of the Thymus to the Radical Resection of Thyroid Cancer and the Protection of Parroid Function
Brief Title: The Importance of Thymus Anatomy to the Radical Resection of Thyroid Cancer Surgery and the Protection of Parathyroid Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20241348
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Thyroid Cancer; Surgery
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thymus anatomy (Experimental): Fine dissection and preservation of thymus tissue are required during surgery.
  Interventions: Procedure: Fine-dissection of the thymus
- non-thymus anatomy (No Intervention): Conventional surgical method for central lymph node dissection

INTERVENTIONS:
Procedure: Fine-dissection of the thymus — In thyroid surgery, precise dissection and preservation of thymus tissue are used to improve the protection of the lower parathyroid gland function and increase the curative effect of the surgery.
  Arms: thymus anatomy

SUMMARY:
Thyroid cancer is one of the most common endocrine malignancies. In the past three decades, the incidence rate of thyroid cancer has continued to rise rapidly in many countries and regions around the world. The incidence rate of thyroid cancer in China is increasing year by year. The standardized incidence rate increased from 1.4/100000 person years in 1990 to 14.65/100000 person years in 2016. It has become the seventh malignant tumor in China with incidence rate, especially the incidence rate of women. Although differentiated thyroid cancer (DTC) has a low degree of malignancy, it still poses a threat to the life, health, and quality of life of patients. Due to its low mortality rate and long survival period, standardized diagnosis, treatment, and follow-up are even more necessary. The 5-year survival rate of thyroid cancer in China has increased significantly from 67.5% in 2003-2005 to 84.3% in 2012-2015, but still lags far behind the 98.3% in the United States.

The current treatment for thyroid cancer is mainly surgical treatment. The development concept of tumor surgery is first radical, followed by functional preservation, and finally aesthetic incision. Standardized and thorough radical surgery is the most critical link to improve patient prognosis and reduce the occurrence of complications. Lymph node metastasis is a common cause of patient recurrence. According to literature reports, the central lymph node metastasis rate after DTC surgery is 24% -64%, which affects the prognosis and quality of life of patients, often requiring secondary surgery, increasing the incidence of postoperative complications and patient burden. Therefore, thyroid cancer surgery requires standardized and thorough neck lymph node dissection. Based on surgical experience and autopsy research, several pre tracheal lymph nodes are often hidden in the deep surface of the thymus from the inferior pole of the thyroid to the upper edge of the unnamed artery. Postoperative recurrence of central lymph nodes often occurs in this area. Therefore, during the initial surgery, the neck segment of the thymus must be freed and pulled away to the shallow layer to thoroughly clean the pre tracheal lymph nodes hidden in the deep surface of the thymus. A considerable number of zone VII lymph nodes can also be pulled out to make the central lymph node cleaning more thorough. However, current surgical standards and guidelines do not emphasize the importance of thymus anatomy.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with thyroid cancer who require total thyroidectomy and bilateral central lymph node dissection.
* The subjects voluntarily joined this study, signed an informed consent form, had good compliance, and cooperated with follow-up.
* Age at the time of signing the informed consent form is between 18 and 80 years old, regardless of gender.
* The physical fitness score of the Eastern Cooperative Oncology Group (ECOG) is 0 or 1.
* Expected survival period is not less than 1 year.
* Male and female patients of childbearing age agreed to use reliable methods of contraception before entering the trial, during the research process, and up to 8 weeks after discontinuation of medication.
* Good organ function:

Hematology: Absolute neutrophil count (ANC) ≥ 1500/μ L; Platelets ≥ 100000/μ L; Hemoglobin ≥ 9.0g/dL or ≥ 5.6 mmol/L; Kidney: Serum creatinine ≤ 1.5 times ULN or calculated creatinine clearance rate (CrCl) ≥ 60 mL/min (using the Cock Gault formula); Liver: For subjects with total bilirubin levels ≤ 1.5 × ULN or for subjects with total bilirubin levels>1.5 × ULN, direct bilirubin is within normal limits; AST (SGOT) and ALT (SGPT) ≤ 2.5 × ULN; Endocrine system: Thyroid stimulating hormone (TSH) is within normal limits. Note: If TSH is not within the normal range at baseline, and if T3 and free T4 are within the normal range, the subject still meets the inclusion criteria; Coagulation function: International normalized ratio (INR) or prothrombin time (PT), activated partial thromboplastin time (aPTT) ≤ 1.5 × ULN, except for subjects undergoing anticoagulant therapy as long as PT or aPTT is within the prescribed range of use of the anticoagulant drug; Willing and able to comply with the visit, treatment plan, laboratory tests, and other research procedures outlined in the research plan.

Exclusion Criteria:

* There are locally advanced unresectable or metastatic diseases.
* History of non infectious pneumonia/interstitial lung disease requiring steroid treatment, or current pneumonia/interstitial lung disease requiring steroid treatment.
* Known history of active tuberculosis.
* Known to have active infections that require systematic treatment.
* Any subjects with known or suspected autoimmune diseases or immune deficiencies.
* Uncontrolled active hepatitis B (defined as hepatitis B B virus surface antigen [HBsAg] test result in screening period is positive and HBV-DNA test value is higher than the upper limit of normal value in the laboratory department of the research center.
* Subjects with HBV-DNA levels<500 IU/mL within 28 days prior to randomization, who have received local standard antiviral treatment for at least 14 days and are willing to continue receiving antiviral treatment during the study period, are eligible for enrollment; Subjects with active hepatitis C (defined as those who test positive for hepatitis C virus surface antibody [HCsAb] and HCV-RNA during the screening period).
* Known human immunodeficiency virus (HIV) infection (known to be HIV antibody positive).
* Administer a live vaccine within 30 days prior to the first dose.
* Have ≥ grade 2 peripheral neuropathy.
* Has experienced severe allergic reactions to other monoclonal antibodies.
* Known to have serious or uncontrolled underlying diseases; Including but not limited to hemodynamic instability cardiovascular events, symptomatic cerebrovascular events, and Child Pugh A or higher liver cirrhosis that occur within 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The effectiveness of surgery | 13 months
  Count the number of central lymph node dissection and positive lymph nodes in routine pathological examination after surgery. Follow up neck ultrasound will be conducted at 3 months, 6 months, and 1 year after surgery, and then every 6 months.

SECONDARY OUTCOMES:
the PTH level after surgery | 13 months
  Dynamic monitoring of PTH changes will be conducted at 1 day, 1 week, 1 month, 3 months, 6 months, and 1 year after surgery until disease progression or recurrence or initiation of new anti-tumor treatment, whichever occurs first.

OTHER OUTCOMES:
Survival situation | 13 months
  The disease-free survival (DFS) evaluated by IRC and researchers is defined as the time from the day of surgery to the first recorded occurrence of local or distant recurrence or death from any cause, whichever occurs first.
  Survival (OS) follow-up: After 30 days of treatment, a 3-month follow-up will be conducted to obtain survival information and subsequent anti-tumor treatment information of the subjects through telephone follow-up or other means, until death, loss to follow-up, withdrawal of informed consent, or termination of the study by the sponsor.